CLINICAL TRIAL: NCT00665782
Title: Stress Measures in Women With Newly Diagnosed Breast Cancer
Brief Title: Measuring Stress in Women With Newly Diagnosed Stage I, Stage II, or Stage III Breast Cancer or Ductal Carcinoma In Situ of the Breast
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00004300; P30CA012197 (NIH); CCCWFU-97307
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Anxiety Disorder; Breast Cancer; Depression; Psychosocial Effects of Cancer and Its Treatment
Keywords: anxiety disorder; depression; psychosocial effects of cancer and its treatment; ductal breast carcinoma in situ; breast cancer in situ; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Depression; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: assessment of therapy complications
Procedure: psychosocial assessment and care
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Gathering information about how patients respond to stress and measuring stress levels in women with newly diagnosed breast cancer may help doctors provide better methods of treatment and on-going care.

PURPOSE: This research study is measuring stress in women with newly diagnosed stage I, stage II, or stage III breast cancer or ductal carcinoma in situ of the breast.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Describe the distributions of physiologic, psychosocial, and behavioral response to stress in women with newly diagnosed breast cancer.
* Describe the patterns of diurnal cortisol rhythms in women newly diagnosed with breast cancer.

Secondary

* Determine if diurnal salivary cortisol (mean or pattern) is consistent over two days within two weeks of study entry.
* Assess the changes in diurnal cortisol rhythm pattern and night-time urinary epinephrine excretion change after an intervening stress event (pre- to post-surgery).
* Determine if the diurnal cortisol rhythm and the night-time urinary excretion correlate with a variety of self-reported psychosocial factors: optimism (LOT-R), state and trait anxiety (STAI form Y-2), positive and negative affect (PANAS), depressive symptoms (CES-D), coping (Brief COPE), and perceived stress (PSS-10).
* Determine if the diurnal cortisol rhythm and the night-time urinary epinephrine excretion correlate with socioeconomic stress and discrimination (functional social support and discrimination [EOD]).
* Determine if the diurnal cortisol rhythm and the night-time urinary epinephrine excretion correlate with one lifestyle behavior and dietary fat consumption (Block food screener).

OUTLINE: Patients are stratified according to race (Caucasian vs African American).

Patients are instructed to collect saliva and urine samples on 2 separate days, within 2 weeks of study enrollment. Saliva samples are collected 6 times a day at baseline, before breast cancer surgery, and 7-10 days after surgery. Urine samples are collected after midnight until and including the first morning sample on the saliva-collection days.

Patients also complete questionnaires (either by telephone interview or in person) within 2 weeks of study enrollment and 7-10 days after breast surgery. Stress measures examined include optimism (LOT-R), trait-anxiety scale (STAI form Y-2), functional social support, affect and depression (PANAS and CES-D), perceived stress (PSS-10), economic hardship scales, discrimination (EOD), coping mechanisms (Brief COPE), and dietary fat consumption (Block Sugar/Fat/Fruit/Vegetable screener).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage I-III invasive breast cancer or ductal carcinoma in situ of the breast within the past 2 weeks
* Surgery for breast cancer planned
* Hormone receptor status not specified
* Female
* Menopausal status not specified
* Able to refrain from:

  * Smoking cigarettes for the 24-hour period of saliva-sample collection
  * Brushing teeth or eating for up to one hour prior to saliva collection
* More than 1 year since prior therapy for another malignancy
* At least 1 month since prior withdrawal from hormone-replacement product
* Able to refrain from steroid inhalers for greater than 24 hours
* No chronic oral steroids

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those diagnosed with stage I-III invasive breast cancer or ductal carcinoma in situ of the breast within the past 2 weeks
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Diurnal cortisol rhythm | Up to 10 days

SECONDARY OUTCOMES:
Consistency of diurnal salivary cortisol levels over two days | Up to 10 days
Changes in diurnal cortisol rhythm pattern and night-time urinary epinephrine excretion pre- to post-surgery | Up to 10 days
Correlation of the diurnal cortisol rhythm and the night-time urinary excretion with the measures of psychosocial and behavioral stress responses | Up to 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Julia A. Lawrence, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States